CLINICAL TRIAL: NCT04819815
Title: Investigation of Chronotropic Response, Exercise Capacity, Quality of Life, Peripheral and Respiratory Muscle Strength in Patients With Type 1 Diabetes Mellitus
Brief Title: Investigation of Chronotropic Index, Exercise Capacity in Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi University 26
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes mellitus; Chronotropic index; Exercise Capacity; Pulmonary Function
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 diabetes mellitus: Patients
  Maximal exercise capacity (Incremental shuttle walk test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), peripheral muscle strength (dynamometer), respiratory muscle endurance ( incremental threshold loading test), physical activity level (multi sensor activity monitor), quality of life (World Health Organization (WHO) well-being index), fatigue (fatigue severity scale), shortness of breath (Modified Medical Research Council MMRC) will be evaluated.
- Healthy Controls: Maximal exercise capacity (Incremental shuttle walk test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), peripheral muscle strength (dynamometer), respiratory muscle endurance ( incremental threshold loading test), physical activity level (multi sensor activity monitor), quality of life (World Health Organization (WHO) well-being index), fatigue ( fatigue severity scale), shortness of breath (Modified Medical Research Council MMRC) will be evaluated.

SUMMARY:
To investigate whether diabetes affects lung function and exercise capacity and impairs autonomic nervous system.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus is a systemic disease that affects the biochemical, morphological and functional properties of various tissues of the body. It is characterized by the loss of insulin-producing cells associated with an autoimmune disorder.

The chronotropic response is an increase in heart rate due to physical activity and metabolic demand. Chronotropic disorder is an inadequate cardiac response and is frequently encountered in individuals with diabetes. Diabetes-related comorbidities or physiological abnormalities may lead to impaired chronotropic response, such as altered blood catecholamine levels during exercise, structural myocardial anomalies, and impaired baroreflex sensitivity. While there are studies on chronotropic response in individuals with type 2 diabetes, chronotropic disorders have not been investigated in adults with type 1 diabetes.

Diabetes affects the lungs negatively. In individuals with diabetes decreased lung volume, and diffusion were observed. Dynamic lung capacity of individuals with type 1 diabetes with the pulmonary function test will be investigated.

There are limited studies evaluating respiratory muscle strength and endurance in individuals with type 1 diabetes. These studies have presented conflicting findings. Informations will be provided to literature by evaluating respiratory muscle strength and endurance.

Physical activity is positively correlated with in the cardiovascular risk factor. Hyperglycemia stresses or fear of hypoglycemia experienced by individuals with type 1 diabetes may lead people to a sedentary life.

Physical activity level of individuals with type 1 diabetes will be evaluated using metabolic holter, which is an objective method.

Patients and healthy individuals will be evaluated and compared. According to the sample size analysis, 27 patients and 27 healthy individuals with similar demographic characteristics will be included in the study. Evaluations will be completed within two days.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients group:

* Individuals aged 18-65 years diagnosed with Type 1 diabetes by basic clinical and laboratory techniques
* Individuals using pump and injection insulin to control type 1 diabetes

Inclusion criteria for healthy group:

* Willing to participate to the study
* Between ages of 18 and 65

Exclusion Criteria:

Exclusion criteria for patients group:

* Individuals with body mass index> 30 kg / m²
* those with lower limb amputation
* those with any heart disease
* Individuals with type 2 diabetes
* Individuals who smoke 10 pack×years
* Anemia
* Individuals with diabetic foot
* Individuals with orthopedic problems
* Individuals with balance problems
* Myocardial infarction or other acute cardiac events within 2 days
* Unstable angina
* Uncontrolled heart rhythm causing symptoms or hemodynamic effects
* Uncontrolled symptomatic heart failure
* Acute pulmonary embolism or pulmonary infarction
* Acute myocarditis or pericarditis
* Suspected or known dissection aneurysm,
* Having an acute systemic infection accompanied by fever, body aches or swollen lymph nodes

Exclusion criteria for healthy group:

* Body mass index> 30 kg / m²
* Smoking exposure 10 pack×years
* Individuals with any chronic illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 27 patients with Type 1 Diabetes mellitus and 27 healthy individuals will be included.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | First Day
  The maximal exercise capacity of the individuals will be evaluated by the incremental shuttle walk test. This test is a symptom-limited maximal field test that evaluates maximal exercise capacity with progressively increased walking speed.
Chronotropic index | First Day
  The chronotropic index will be calculated using the results of the maximal exercise test.

SECONDARY OUTCOMES:
Pulmonary function (Forced vital capacity (FVC)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (FEV1 / FVC) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, peak flow rate (PEF) will be evaluated.
Respiratory Muscle Strength | Second Day
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device.
Respiratory Muscle Endurance | Second Day
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd. Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load.
  The test will be started with 20% of the maximal inspiratory pressure and the pressure will be increased to 40%, 60%, 80%, and 100% every two minutes. Patients will be asked to continue breathing through the device during the test. During the test, the number of breaths delivered during each 2-minute period will be recorded. If the individual cannot breathe 3 consecutive times, the test will be terminated by the physiotherapist.
  The total duration of the test and the maximum pressure value at which it continues to breathe for at least 1 minute will be multiplied. The value found will be recorded as the respiratory muscle endurance value.
Peripheral Muscle Strength | Second Day
  Knee extensor muscle strength using portable hand held dynamometer will be evaluated.
Physical Activity Level | Second Day
  Physical activity will be evaluated multi sensor activity monitor.
Shortness of breath | First Day
  The Modified Medical Research Council (MMRC) dyspnea scale will be used to determine dyspnea perception during daily living activities.
  Dyspnea is graded as: zero (shortness of breath with strenuous exercise only); one (shortness of breath when rushing or walking up a slight uphill); two (because of shortness of breath they walk slower than people of the same age or have to stop to breathe while walking at their own pace); three (stops to breathe after walking 100 meters or after a few minutes); and four (too short of breath to leave the house or shortness of breath when getting dressed).
Fatigue | First Day
  Fatigue will be evaluated using Turkish version of Fatigue Severity Scale. This questionnaire includes 9 items and score range for each item from 1 to 7 point (7-point Likert scale). Fatigue Severity Scale score is calculates by deriving an arithmetic mean. Cut-scores of over 4 are indicative of significant fatigue (higher scores show more severe fatigue).
Life Quality | First Day
  It will be evaluated by Turkish adaptation of the World Health Organization (WHO) well-being index.

CONTACTS AND LOCATIONS:
Overall Officials: Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi Universitiy; Ayşenur SARISAKALOĞLU, Pt, Study Chair — Gazi Universitiy; Meriç COŞKUN, Dr., Principal Investigator — Gazi Universitiy; Füsun BALOŞ TÖRÜNER, Prof.Dr., Principal Investigator — Gazi Universitiy
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sydo N, Sydo T, Merkely B, Carta KG, Murphy JG, Lopez-Jimenez F, Allison TG. Impaired Heart Rate Response to Exercise in Diabetes and Its Long-term Significance. Mayo Clin Proc. 2016 Feb;91(2):157-65. doi: 10.1016/j.mayocp.2015.10.028. Epub 2016 Jan 5. PMID 26769183
- [Background] Komatsu WR, Gabbay MA, Castro ML, Saraiva GL, Chacra AR, de Barros Neto TL, Dib SA. Aerobic exercise capacity in normal adolescents and those with type 1 diabetes mellitus. Pediatr Diabetes. 2005 Sep;6(3):145-9. doi: 10.1111/j.1399-543X.2005.00120.x. PMID 16109070
- [Background] Goldman MD. Lung dysfunction in diabetes. Diabetes Care. 2003 Jun;26(6):1915-8. doi: 10.2337/diacare.26.6.1915. No abstract available. PMID 12766133
- [Background] Fuso L, Pitocco D, Longobardi A, Zaccardi F, Contu C, Pozzuto C, Basso S, Varone F, Ghirlanda G, Antonelli Incalzi R. Reduced respiratory muscle strength and endurance in type 2 diabetes mellitus. Diabetes Metab Res Rev. 2012 May;28(4):370-5. doi: 10.1002/dmrr.2284. PMID 22271438
- [Background] Miculis CP, De Campos W, da Silva Boguszweski MC. Correlation between glycemic control and physical activity level in adolescents and children with type 1 diabetes. J Phys Act Health. 2015 Feb;12(2):232-7. doi: 10.1123/jpah.2013-0024. Epub 2014 Feb 5. PMID 24508755